CLINICAL TRIAL: NCT03558334
Title: Intravenous Human Umbilical-Cord-Derived Mesenchymal Stem Cells For Moderate and Severe Bronchopulmonary Dysplasia in Premature Infants
Brief Title: Human Mesenchymal Stem Cells For Bronchopulmonary Dysplasia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xia Yunqiu, doctor, Children's Hospital of Chongqing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XYunqiu
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary Dysplasia; human umbilical cord -derived mesenchymal stem cells
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transplantation of Mesenchymal Stem Cell (Experimental): Mesenchymal stem cell will be given to preterm infants with BPD.
  Interventions: Drug: Transplantation of mesenchymal stem cell
- No Transplantation of Mesenchymal Stem Cell (Active Comparator): Mesenchymal stem cell will be not given to preterm infants with BPD.
  Interventions: Drug: No transplantation of mesenchymal stem cell

INTERVENTIONS:
Drug: Transplantation of mesenchymal stem cell — Human umbilical cord-derived mesenchymal stem cell will be given to preterm infants through intravenous infusion.
  Dose A - 1 million cells per kg Dose B - 5 million cells per kg
  Other Names: Intravenous infusion of mesenchymal stem cell
  Arms: Transplantation of Mesenchymal Stem Cell
Drug: No transplantation of mesenchymal stem cell — Human umbilical cord-derived mesenchymal stem cell will be not given to preterm infants through intravenous infusion.
  Other Names: No intravenous infusion of mesenchymal stem cell
  Arms: No Transplantation of Mesenchymal Stem Cell

SUMMARY:
This study is an open-label, single-center, dose escalation study to evaluate of safety and efficacy of human umbilical cord -derived mesenchymal stem cells (hUC-MSCs) in premature infants for moderate and severe Bronchopulmonary Dysplasia（BPD）.

DETAILED DESCRIPTION:
BPD is a chronic lung disease that occur in premature infants receiving prolonged oxygen pulmonary and ventilator therapy. It remains a main complication of extreme prematurity and currently lacks efficient treatment.The mortality rate of one year after birth is still high and the quality of life is not optimistic.

hUC-MSCs are widely used in clinic due to their low immunogenicity and convenient to get.Many animal study had shown that hUC-MSCs had therapeutic effects on a variety of animal models of lung disease.Furthermore,there are a large number of clinical trials of MSCs applied to various system diseases and the safety was verified.So,the main purpose of this study is to evaluate the safety and efficacy of hUC-MSCs in participants with moderate and severe BPD.

ELIGIBILITY:
Inclusion Criteria:

1. The participants meet the diagnostic criteria for moderate and severe BPD established by the National Institutes of Child Health and Human Development (NICHD) workshop.
2. The participants have abnormal respiratory manifestations.
3. Written consent form signed by a legal representative or a parent.

Exclusion Criteria:

1. Although mechanical ventilation or oxygen is required in participants, there are no signs of dyspnea or BPD-related changes in lung imaging, such as central apnea or diaphragm paralysis.
2. The participants who have complex congenital heart disease.
3. The participants who have severe pulmonary hypertension(cardiac ultrasound confirmed) at the time of assessment.
4. The participants who have severe respiratory tract malformation: pierre-robin syndrome, tracheobronchomalacia, vascular ring syndrome, congenital tracheal stenosis, tracheo-esophageal fistula, pulmonary emphysema, pulmonary sequestration, congenital pulmonary dysplasia, congenital pulmonary cyst, congenital spasm, etc.
5. The participants who have severe chromosome anomalies :Edward syndrome, Patau syndrome, Down syndrome, etc) or severe congenital malformation (Hydrocephalus, Encephalocele, etc).
6. The participants who have severe congenital infection(Herpes, Toxoplasmosis, Rubella, Syphilis, AIDS, etc).
7. The participants who have severe sepsis or shock.
8. The participants who is going to have surgery 72 hours before/after this study drug administration.
9. The participants who have surfactant administration within 24 hours before this study drug administration.
10. The participants who have severe intracranial hemorrhage ≥ grade 3 or 4.
11. The participants who have active pulmonary hemorrhage or active air leak syndrome at the time of assessment.
12. The participants who have the history of other clinical studies as a participant.
13. The participants who is considered inappropriate by the investigators.

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-06-28 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse reactions related to infusion after treatment | 24 hours after administration
  To evaluate the safety of human umbilical cord -derived mesenchymal stem cells for BPD.

SECONDARY OUTCOMES:
Changes of high-resolution chest CT in participants | within 2 years after administration
  To evaluate the safety and efficacy of human umbilical cord -derived mesenchymal stem cells for BPD.
Changes of temperature in participants | 3 days after administration
  To evaluate the safety of human umbilical cord -derived mesenchymal stem cells for BPD.
Changes of blood pressure in participants | 3 days after administration
  To evaluate the safety of human umbilical cord -derived mesenchymal stem cells for BPD. Blood pressure is measured by electronic sphygmomanometer .
Changes of heart rate in participants | 3 days after administration
  To evaluate the safety of human umbilical cord -derived mesenchymal stem cells for BPD.
Changes of respiratory rate in participants | 3 days after administration
  To evaluate the safety of human umbilical cord -derived mesenchymal stem cells for BPD.
Changes of oxygen saturation in participants | 3 days after administration
  To evaluate the safety of human umbilical cord -derived mesenchymal stem cells for BPD.
Growth velocity (Z-score) in participants | within 2 years after administration
  To evaluate the safety and efficacy of human umbilical cord -derived mesenchymal stem cells for BPD.

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Fu, Study Chair — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang YS, Ahn SY, Yoo HS, Sung SI, Choi SJ, Oh WI, Park WS. Mesenchymal stem cells for bronchopulmonary dysplasia: phase 1 dose-escalation clinical trial. J Pediatr. 2014 May;164(5):966-972.e6. doi: 10.1016/j.jpeds.2013.12.011. Epub 2014 Feb 6. PMID 24508444
- [Background] Hayes D Jr, Meadows JT Jr, Murphy BS, Feola DJ, Shook LA, Ballard HO. Pulmonary function outcomes in bronchopulmonary dysplasia through childhood and into adulthood: implications for primary care. Prim Care Respir J. 2011 Jun;20(2):128-33. doi: 10.4104/pcrj.2011.00002. PMID 21336467
- [Background] Ahn SY, Chang YS, Kim JH, Sung SI, Park WS. Two-Year Follow-Up Outcomes of Premature Infants Enrolled in the Phase I Trial of Mesenchymal Stem Cells Transplantation for Bronchopulmonary Dysplasia. J Pediatr. 2017 Jun;185:49-54.e2. doi: 10.1016/j.jpeds.2017.02.061. Epub 2017 Mar 21. PMID 28341525
- [Background] Wilson JG, Liu KD, Zhuo H, Caballero L, McMillan M, Fang X, Cosgrove K, Vojnik R, Calfee CS, Lee JW, Rogers AJ, Levitt J, Wiener-Kronish J, Bajwa EK, Leavitt A, McKenna D, Thompson BT, Matthay MA. Mesenchymal stem (stromal) cells for treatment of ARDS: a phase 1 clinical trial. Lancet Respir Med. 2015 Jan;3(1):24-32. doi: 10.1016/S2213-2600(14)70291-7. Epub 2014 Dec 17. PMID 25529339
- [Background] Laube M, Stolzing A, Thome UH, Fabian C. Therapeutic potential of mesenchymal stem cells for pulmonary complications associated with preterm birth. Int J Biochem Cell Biol. 2016 May;74:18-32. doi: 10.1016/j.biocel.2016.02.023. Epub 2016 Feb 27. PMID 26928452
- [Background] Pierro M, Ionescu L, Montemurro T, Vadivel A, Weissmann G, Oudit G, Emery D, Bodiga S, Eaton F, Peault B, Mosca F, Lazzari L, Thebaud B. Short-term, long-term and paracrine effect of human umbilical cord-derived stem cells in lung injury prevention and repair in experimental bronchopulmonary dysplasia. Thorax. 2013 May;68(5):475-84. doi: 10.1136/thoraxjnl-2012-202323. Epub 2012 Dec 4. PMID 23212278
- [Background] Hansmann G, Fernandez-Gonzalez A, Aslam M, Vitali SH, Martin T, Mitsialis SA, Kourembanas S. Mesenchymal stem cell-mediated reversal of bronchopulmonary dysplasia and associated pulmonary hypertension. Pulm Circ. 2012 Apr-Jun;2(2):170-81. doi: 10.4103/2045-8932.97603. PMID 22837858
- [Derived] Xia Y, Lang T, Niu Y, Wu X, Zhou O, Dai J, Bao L, Yang K, Zou L, Fu Z, Geng G. Phase I trial of human umbilical cord-derived mesenchymal stem cells for treatment of severe bronchopulmonary dysplasia. Genes Dis. 2022 Feb 22;10(2):521-530. doi: 10.1016/j.gendis.2022.02.001. eCollection 2023 Mar. PMID 37223507